CLINICAL TRIAL: NCT04221087
Title: Dexamethasone Use for the Treatment of Non-RSV Bronchiolitis
Brief Title: Steroid Use in Non-RSV Bronchiolitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID19-pandemic, RSV surge
Sponsor: Allison Williams (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor-Investigator, Allison Williams, Assistant Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19080287
Record Dates: First submitted 2019-12-29; First posted 2020-01-09 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Bronchiolitis, Viral
Keywords: bronchiolitis; non-RSV bronchiolitis; dexamethasone; treatment; steroid
MeSH Terms: conditions — Bronchiolitis, Viral; Bronchiolitis | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either intervention or control group upon admission if they meet inclusion/exclusion criteria and consent.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Arm (Placebo Comparator): Participants will be given a placebo of sugar water (0.6ml/kg/dose) in a single oral dose and standard of care for bronchiolitis (supplemental oxygen, antipyretics, suctioning etc.)
  Interventions: Drug: Placebos
- Dexamethasone Arm (Experimental): Participants will be given dexamethasone (0.6mg/kg/dose) in a single oral dose in addition to the standard of care for bronchiolitis (supplemental oxygen, antipyretics, suctioning etc.)
  Interventions: Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Placebos — Sugar water based on same ml dosing of intervention arm drug
  Other Names: sugar water
  Arms: Placebo Arm
Drug: Dexamethasone Oral — 0.6mg/kg/dose - single oral dose administration to intervention arm
  Other Names: Decadron
  Arms: Dexamethasone Arm

SUMMARY:
The proposed study is a pilot randomized control trial to determine the efficacy of dexamethasone use in hospitalized children who are less than 2 years of age with non-respiratory syncytial virus (RSV) bronchiolitis admitted to the University of Pittsburgh Medical Center (UPMC) Children's Hospital of Pittsburgh from February 1 to May 31, 2022. It is hypothesized that the use of standard airway-dose steroids (0.6mg/kg dexamethasone) will improve the clinical outcome of children hospitalized for non-RSV bronchiolitis, which will be evident by decreased length of stay.

DETAILED DESCRIPTION:
The study will take place at UPMC Children's Hospital of Pittsburgh with patients admitted to the general pediatric service. The attending physician on the clinical service team will identify patients diagnosed with bronchiolitis. If the participant meets inclusion and exclusion criteria, a member from the study team will then meet with the participant's family to discuss the study and obtained informed consent. A participant may have had a rapid RSV/influenza testing already complete for clinical purposes. If this has been done, participants will be asked to obtain a secondary nasopharyngeal swab so that it may be tested for a full respiratory viral panel for statistical stratification. Once rapid testing is obtained and results are negative for both RSV and influenza, the participant will then be randomized to either the intervention (dexamethasone) or control (placebo) arm of the study. Study members will calculate a modified Tal score (MTS) at time of consent and then 12-24 hours after medication administration. Throughout admission, participants will also receive standard of care for bronchiolitis, which may include regular vital sign evaluation, supplemental oxygen, intravenous fluids or nasogastric tube feedings, and anti-pyretic therapy. Because this is a pilot study, the study will be underpowered, however, this study will provide data that will allow the investigators to estimate the sample size needed for a future study. The number of time points to be used for the generalized estimating equation can be determined ad hoc to include a reasonably balanced sample to make the comparison valid.

ELIGIBILITY:
Inclusion Criteria:

1. Less than or equal to 24 months
2. First episode of wheezing or first clinical diagnosis of bronchiolitis
3. Admitted to the general pediatric service at UPMC Children's Hospital of Pittsburgh
4. Ability of a parent or guardian to understand and comply with the study procedures
5. Signed written informed consent by parent or guardian

Exclusion Criteria:

1. Preterm birth < 35 weeks
2. Presence of underlying cardiopulmonary, neuromuscular, or other complex disease
3. Admission to the pediatric intensive care unit
4. Co-infection with influenza infection or concomitant bacterial infection (such as pneumonia or AOM)
5. History of allergy or reaction to steroids
6. History of an underlying chronic medical condition -including chronic heart disease, chronic lung disease (except asthma),congenital anomalies of the airways or lung, cystic fibrosis, chronic renal disease including nephrotic syndrome, protein losing enteropathy of any cause, severe malnutrition, neurocognitive disorders, metabolic disorders (including phenylketonuria), or genetic disorders (note: genetic syndromes such as Down syndrome and Edwards Syndrome are excluded; however, children with genetic disorders (e.g., hemophilia) but who do not have a genetic syndrome may not satisfy this particular exclusion criterion; it is important that children with such genetic disorders do not have symptoms and/or comorbidities that would pose additional risk to them nor jeopardize the adequacy of study assessments.")
7. History of a condition that compromises the immune system - human immunodeficiency virus infection, primary immunodeficiency, anatomic or functional asplenia; receipt of a hematopoietic stem cell or solid organ transplant at any time; receipt of immunosuppressive therapy including chemotherapeutic agents, biologic agents, antimetabolites or radiation therapy during the past 12 months; or daily use of systemic corticosteroids for more than 7 consecutive days during the past 14 days.
8. Any other condition that in the judgment of the investigator precludes participation because it could affect the safety of the subject

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison E Williams, MD, Principal Investigator — University of Pittsbrgh, UPMC Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Arm | Dexamethasone Arm
Started | 2 | 1
Completed | 2 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Dexamethasone Arm | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: months] | 2.75 (1.77) | 12 (NA) — only one participant | 5.83 (5.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Measurement of hospital length of stay in hours
Time Frame: Admission vitals through discharge paperwork printing time, average of 24-96 hours
Population: No data was collected
Arm/Group | Placebo Arm | Dexamethasone Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Severity of Bronchiolitis
Description: Measurement of reducing severity of bronchiolitis by assessment with modified TAL score (MTS)
Time Frame: Will obtain MTS upon admission by chart view or, if unable, at time of enrollment, and compare to MTS obtained 12 hours after medication administration
Population: No data was collected
Arm/Group | Placebo Arm | Dexamethasone Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Severity of Bronchiolitis
Description: Measurement of reducing severity of bronchiolitis by assessment with modified TAL score (MTS)
Time Frame: Will compare respiratory assessment via MTS 12 hours after admission and at discharge, average of 24-96 hours from admission
Population: No data was collected
Arm/Group | Placebo Arm | Dexamethasone Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Severity of Bronchiolitis
Description: Measurement of reducing severity of bronchiolitis by evaluation of patient outcome - discharge, transfer to ICU or acute care floor
Time Frame: Admission to time of discharge to home or transfer to ICU or acute care floor, usual time frame is 24-72 hours
Population: No data was collected
Arm/Group | Placebo Arm | Dexamethasone Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: 7-day Same-Cause Revisit Rate
Description: Measuring number of revisits to the primary care physician or emergency room or re-admission to the hospital for ongoing bronchiolitis related symptoms within 7 days of discharge
Time Frame: Discharge to 7 days
Population: No data was collected
Arm/Group | Placebo Arm | Dexamethasone Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12-36 hours (length of hospital admission)
Groups:
- Placebo: Participants will be given a placebo of sugar water (0.6ml/kg/dose) in a single oral dose and standard of care for bronchiolitis (supplemental oxygen, antipyretics, suctioning etc.)
- Dexamethasone: Participants will be given dexamethasone (0.6mg/kg/dose) in a single oral dose in addition to the standard of care for bronchiolitis (supplemental oxygen, antipyretics, suctioning etc.)
Arm/Group | Placebo | Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT04221087/Prot_SAP_000.pdf